CLINICAL TRIAL: NCT06068764
Title: Etomidate Versus Propofol As An Anesthesia Induction Agent For Patients Undergoing CABG Surgery, Assessing Hemodynamic Stability. A Single Blinded, Randomized Controlled Trial.
Brief Title: Etomidate Versus Propofol in CABG Surgery
Acronym: ETOPRO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Joseph Hinchey, Principal Investigator, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HHC-2023-0114
Record Dates: First submitted 2023-08-10; First posted 2023-10-05 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease
Keywords: CABG surgery; Etomidate; Propofol; general anesthesia induction agenats; cardiothoracic anesthesia
MeSH Terms: conditions — Coronary Artery Disease | interventions — Etomidate; Propofol

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, single-blinded, randomized controlled clinical trial
Who Masked: Participant
Masking Description: Due to the difference in the physical appearance of etomidate and propofol medications, the anesthesiologist administering any of these medications will not be blinded. Only study patients will be blinded to the anesthesia induction agent they receive. Therefore, this study is considered single-blinded.
  Since this is a clinical trial, blinding is an important method to reduce bias and ensure the validity of study results. Unblinding is unnecessary in this study unless the situation when a participant experiences a serious adverse event that is unexpected and related to the anesthesia induction agent (study intervention) and the course of treatment needs to be adjusted. Unblinding in this situation will be the decision of the principal investigator (PI). The PI will unblind the patient (i.e., tell the patient about the assigned group), and take any additional necessary course of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Etomidate (Experimental): Etomidate as the principal hypnotic agent in a single bolus dose of 0.2-0.3 mg/kg along with 250mcg of fentanyl, 50mg ketamine, 0.7 mg/kg rocuronium, and 5ml of 2% lidocaine.
  Interventions: Drug: Etomidate
- Propofol (Active Comparator): Propofol as the principal hypnotic agent in a single bolus dose of 50mg of propofol along with 250 mcg of fentanyl, 50mg ketamine, 0.7 mg/kg rocuronium, and 5ml of 2% lidocaine.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Etomidate — The type of general anesthesia induction agent for CABG surgery
  Other Names: Amidate™
  Arms: Etomidate
Drug: Propofol — The type of general anesthesia induction agent for CABG surgery
  Other Names: Diprivan
  Arms: Propofol

SUMMARY:
The objective of this single-blinded randomized controlled interventional clinical trial is to learn about the efficacy and long-term safety of etomidate compared to propofol as an anesthesia induction agent in patients undergoing coronary artery bypass graft (CABG) surgery. The primary aim of this study is to determine whether patients receiving etomidate or propofol exhibit similar requirements for vasopressor or ionotropic agents during both the intraoperative and postoperative periods.

To achieve this goal, participants who are scheduled for CABG surgery will be randomly assigned to receive either etomidate or propofol as the principal hypnotic agent. The researchers will then compare the effects of these two anesthesia induction agents on various factors, including the need for hemodynamic support, hemodynamic stability, duration of mechanical ventilation, length of stay in the intensive care unit (ICU), and overall hospital length of stay. Additionally, they will assess whether there are disparities in mortality rates and readmission rates within a 6-month timeframe after the surgery.

By comparing the outcomes between the two groups, the study aims to provide valuable insights into the potential differences in vasopressor or ionotropic agent requirements between etomidate and propofol. This information can help inform clinical decision-making and potentially optimize anesthesia management strategies for patients undergoing CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for elective open coronary arteries bypass graft CABG surgery
2. Patients with American Society of Anesthesiology (ASA) physical status score I- IV
3. Patients with the ability to speak and read both English and Spanish

Exclusion Criteria:

1. Emergency CABG surgery, STAT cases, and add-on cases.
2. Refusal or lack of providing the study consent
3. Patients with a known current adrenocortical insufficiency
4. A patient who is presenting with any kind of shock, (e.g. septic, hypovolemic, cardiogenic, etc.)
5. Patients with chronic steroid use (defined as the use of glucocorticoids within 6 months preoperatively)
6. Patients with a known allergy to etomidate or propofol.
7. Patients with a known seizure disorder.
8. Patients who are enrolled in other clinical research studies that can compete with this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Vasopressors dose expressed by Noradrenaline Equivalent dose [μg/kg/min] | 30 minutes after induction, last 30 minutes of post bypass period, and first 24 hours post procedure.
  Vasopressor requirements will be expressed as Noradrenaline Equivalent dose using the formula of (NEq [μg/kg/min] = norepinephrine + epinephrine + phenylephrine/10 + dopamine/100 + vasopressin*2.5), this will be measured during three periods of time: Intraoperatively during the first 30 minutes post induction (as a reflection of the impact of induction on hemodynamics), intraoperatively during the last 30 minutes of the post bypass period, and for the first 24 hours post procedure.

SECONDARY OUTCOMES:
The number of incidences of shock | First 24 hours post anesthesia
  The incidence of both vasogenic and cardiogenic shocks will be determined intraoperatively and postoperatively using the Mean Arterial Pressure (MAP), Central Venous Pressure (CVP), Cardiac Output (CO), and Systemic Vascular Resistance (SVR).
  Vasogenic shock (defined as a MAP < 60 mmHg with normal CO (>2.0 L/min) and low SVR (< 900 dynes/sec).
  Cardiogenic shock (defined as hypotension with MAP < 60 mmHg, low CO (<2.0 L/min), and normal SVR range (900-1400 dynes/sec).
ICU length of stay | 3 days
  ICU length of stay will be calculated in hours using the ICU data from EPIC.
Hospital length of stay | 7 days
  Hospital length of stay will be calculated in hours from the date and time of admission and discharge, from EPIC.
Hospital Readmissions | 6 months
  In the 6th month after surgery, a retrospective safety checkup will be done, using EPIC chart review, to assess the number of readmissions.
Time to extubation and end of mechanical ventilation | until extubation, assessed as 6 hours
  Time to extubation, the standard of care is usually within 6 hours of arriving to the unit.
Incidence of Death | 6 months
  In the 6th month after surgery, a retrospective safety checkup will be done, using EPIC chart review, to assess the number of deaths if any.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Hinchey, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hildreth AN, Mejia VA, Maxwell RA, Smith PW, Dart BW, Barker DE. Adrenal suppression following a single dose of etomidate for rapid sequence induction: a prospective randomized study. J Trauma. 2008 Sep;65(3):573-9. doi: 10.1097/TA.0b013e31818255e8. PMID 18784570
- [Background] De Jong A, Jaber S. Etomidate for anesthesia induction: friends or foe in major cardiac surgery? Crit Care. 2014 Oct 10;18(5):560. doi: 10.1186/s13054-014-0560-7. PMID 25672223
- [Background] Ledingham IM, Watt I. Influence of sedation on mortality in critically ill multiple trauma patients. Lancet. 1983 Jun 4;1(8336):1270. doi: 10.1016/s0140-6736(83)92712-5. No abstract available. PMID 6134053
- [Background] Chan CM, Mitchell AL, Shorr AF. Etomidate is associated with mortality and adrenal insufficiency in sepsis: a meta-analysis*. Crit Care Med. 2012 Nov;40(11):2945-53. doi: 10.1097/CCM.0b013e31825fec26. PMID 22971586
- [Background] Erdoes G, Basciani RM, Eberle B. Etomidate--a review of robust evidence for its use in various clinical scenarios. Acta Anaesthesiol Scand. 2014 Apr;58(4):380-9. doi: 10.1111/aas.12289. Epub 2014 Mar 3. PMID 24588359
- [Background] Jabre P, Combes X, Lapostolle F, Dhaouadi M, Ricard-Hibon A, Vivien B, Bertrand L, Beltramini A, Gamand P, Albizzati S, Perdrizet D, Lebail G, Chollet-Xemard C, Maxime V, Brun-Buisson C, Lefrant JY, Bollaert PE, Megarbane B, Ricard JD, Anguel N, Vicaut E, Adnet F; KETASED Collaborative Study Group. Etomidate versus ketamine for rapid sequence intubation in acutely ill patients: a multicentre randomised controlled trial. Lancet. 2009 Jul 25;374(9686):293-300. doi: 10.1016/S0140-6736(09)60949-1. Epub 2009 Jul 1. PMID 19573904
- [Background] McPhee LC, Badawi O, Fraser GL, Lerwick PA, Riker RR, Zuckerman IH, Franey C, Seder DB. Single-dose etomidate is not associated with increased mortality in ICU patients with sepsis: analysis of a large electronic ICU database. Crit Care Med. 2013 Mar;41(3):774-83. doi: 10.1097/CCM.0b013e318274190d. PMID 23318491
- [Background] Hohl CM, Kelly-Smith CH, Yeung TC, Sweet DD, Doyle-Waters MM, Schulzer M. The effect of a bolus dose of etomidate on cortisol levels, mortality, and health services utilization: a systematic review. Ann Emerg Med. 2010 Aug;56(2):105-13.e5. doi: 10.1016/j.annemergmed.2010.01.030. Epub 2010 Mar 25. PMID 20346542
- [Background] Wagner CE, Bick JS, Johnson D, Ahmad R, Han X, Ehrenfeld JM, Schildcrout JS, Pretorius M. Etomidate use and postoperative outcomes among cardiac surgery patients. Anesthesiology. 2014 Mar;120(3):579-89. doi: 10.1097/ALN.0000000000000087. PMID 24296761
- [Background] Heinrich S, Schmidt J, Ackermann A, Moritz A, Harig F, Castellanos I. Comparison of clinical outcome variables in patients with and without etomidate-facilitated anesthesia induction ahead of major cardiac surgery: a retrospective analysis. Crit Care. 2014 Jul 11;18(4):R150. doi: 10.1186/cc13988. PMID 25015112
- [Background] Basciani RM, Rindlisbacher A, Begert E, Brander L, Jakob SM, Etter R, Carrel T, Eberle B. Anaesthetic induction with etomidate in cardiac surgery: A randomised controlled trial. Eur J Anaesthesiol. 2016 Jun;33(6):417-24. doi: 10.1097/EJA.0000000000000434. PMID 26914224
- [Background] Morel J, Salard M, Castelain C, Bayon MC, Lambert P, Vola M, Auboyer C, Molliex S. Haemodynamic consequences of etomidate administration in elective cardiac surgery: a randomized double-blinded study. Br J Anaesth. 2011 Oct;107(4):503-9. doi: 10.1093/bja/aer169. Epub 2011 Jun 17. PMID 21685487
- [Background] Iribarren JL, Jimenez JJ, Hernandez D, Lorenzo L, Brouard M, Milena A, Mora ML, Martinez R. Relative adrenal insufficiency and hemodynamic status in cardiopulmonary bypass surgery patients. A prospective cohort study. J Cardiothorac Surg. 2010 Apr 19;5:26. doi: 10.1186/1749-8090-5-26. PMID 20403156
- [Background] Hannam JA, Mitchell SJ, Cumin D, Frampton C, Merry AF, Moore MR, Kruger CJ. Haemodynamic profiles of etomidate vs propofol for induction of anaesthesia: a randomised controlled trial in patients undergoing cardiac surgery. Br J Anaesth. 2019 Feb;122(2):198-205. doi: 10.1016/j.bja.2018.09.027. Epub 2018 Nov 15. PMID 30686305
- [Background] Goradia S, Sardaneh AA, Narayan SW, Penm J, Patanwala AE. Vasopressor dose equivalence: A scoping review and suggested formula. J Crit Care. 2021 Feb;61:233-240. doi: 10.1016/j.jcrc.2020.11.002. Epub 2020 Nov 14. PMID 33220576